CLINICAL TRIAL: NCT04181593
Title: A Randomized, Multicenter, Double-Masked, Placebo Controlled Study of the Safety and Efficacy of OmegaD Softgels in the Treatment of Dry Eye Disease
Brief Title: Phase 3 Study of the Safety and Efficacy of OmegaD Softgels in the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OmegaD LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OmegaD-2019-002
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye
Keywords: Dry Eye Disease; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OmegaD (Experimental): OmegaD Softgels
  Interventions: Drug: Omega 3 fatty acid
- Placebo (Placebo Comparator): Placebo Softgels
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Omega 3 fatty acid — Omega 3 fatty acid Softgels
  Other Names: OmegaD Softgels
  Arms: OmegaD
Drug: Placebos — Mineral oil Softgels
  Other Names: Placebo Softgels
  Arms: Placebo

SUMMARY:
This is a phase 3 study to evaluate the safety and efficacy of OmegaD softgels for the treatment of dry eye disease. A daily dose of 2 OmegaD softgels dosed orally BID will be compared to 2 placebo softgels (mineral oil ) dosed orally BID for 84 days. Approximately 300 subjects will be evaluated for their signs and symptoms of dry eye disease and for safety throughout the study.

DETAILED DESCRIPTION:
Inflammation is a key component of dry eye disease. Increasing the systemic levels of omega-3 fatty acids relative to omega-6 levels can mediate immune responses. Evaluating whether omega-3 supplementation can improve dry eye disease signs, symptoms and associated measures of inflammation may present a new therapeutic option for dry eye disease.

The primary objective of this study is to evaluate the safety and efficacy of twice daily (BID) dosing of OmegaD softgels in subjects with dry eye disease.

Male and female subjects between 18 years and 90 years of age, with at least moderate ocular surface disease (OSDI ≥ 20) dry eye symptoms and a clinical diagnosis of dry eye disease supported by global clinical assessment will be screened and enrolled. Each subject must have, in at least one eye, tear osmolarity of ≥ 312 mOsm/L and meibomian gland dysfunction as defined by a grade of 1 or 2 on the meibomian orifice size scale at both Screening and Baseline in at least one eye. In addition, Tear break up time (TBUT) must be ≤ 7 seconds in both eyes at Screening and the Schirmer's test score in both eye(s) must be ≥ 5 mm at Screening.

Approximately 300 subjects will be randomized (1:1) to 1 of 2 treatment arms and treated for 84 days (12 weeks) with either OmegaD softgels; 2 softgels BID or placebo softgels; 2 softgels BID. The study will be double-masked with OmegaD and placebo being identical-appearing softgels.

Subjects will participate in safety and efficacy assessments throughout the study. Efficacy assessments will include, tear osmolarity, meibomian gland dysfunction grading, TBUT, Schirmer's Test, and dry eye symptoms based on the OSDI questionnaire, Safety assessments will include, slit lamp examination and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≥ 18 years and ≤ 90 years on the date of informed consent.
2. All subjects must provide signed written consent prior to participation in any study-related procedures.
3. At least moderate ocular surface disease as measured by an OSDI score ≥ 20 at Screening.
4. Clinical diagnosis of dry eye disease supported by global clinical assessment.
5. Presence of tear osmolarity in at least one eye ≥ 312 mOsm/L at both Screening and Baseline.
6. Schirmer's test score (anesthetized) ≥ 5 mm in both eyes at Screening.
7. TBUT ≤ 7 seconds in both eyes at Screening.
8. Presence of meibomian gland dysfunction as defined by a grade of 1 or 2 on the meibomian orifice size scale in at least one eye at both Screening and Baseline. The qualifying osmolarity level and meibomian orifice size grade must be present in the same eye at both Screening and Baseline if only one eye qualifies.

Exclusion Criteria:

1. Any previous reconstructive or cosmetic eyelid surgery that may, in the Investigator's opinion, affect the normal function of the lids (eg, blepharoplasty, ptosis repair, entropion/ectropion repair) that could affect study parameters/assessments.
2. Cataract extraction, with or without minimally invasive glaucoma surgery (eg, iStent), within 90 days prior to Screening.
3. Any previous invasive glaucoma surgery (eg, trabeculectomy, shunts, valves) and/or corneal surgery (eg, penetrating keratoplasty, lamellar keratoplasty, Descemet's stripping endothelial keratoplasty [DSEK]).
4. Lid scrubs with over-the-counter (OTC) products (eg, OCuSOFT lid scrub, SteriLid, baby shampoo, etc.) and/or warm compresses within 14 days prior to Screening and throughout the study period.
5. Prescription and OTC ophthalmic mast cell stabilizers and antihistamines within 21 days prior to Screening and throughout the study period (systemic mast cell stabilizers are allowed, and systemic antihistamines are permitted with certain restrictions [see exclusion criterion 16]).
6. Chronic daily use (defined as > 7 consecutive days at the recommended dosing frequency) of systemic narcotics for any chronic pain syndrome (eg, fibromyalgia, rheumatoid arthritis, etc.) during the study period. Short-term, as-needed dosing of a systemic narcotic for ≤ 72 hours is allowed, but not at Screening or on the day of the study visit.
7. Allergy to fish oil or mineral oil (component of placebo softgels) or any component of the softgel material.
8. Clinically significant eyelid deformity or eyelid movement disorder that is caused by conditions such as notch deformity, incomplete lid closure, entropion, ectropion, hordeolum, or chalazion.
9. Active or anticipated seasonal and/or perennial allergic conjunctivitis or rhinitis.
10. Previous ocular disease leaving sequelae or requiring current topical eye therapy other than for dry eye disease, including, but not limited to, active corneal or conjunctival infection or inflammation of the eye and ocular surface scarring.
11. History or presence of abnormal nasolacrimal drainage.
12. Laser-assisted in situ keratomileusis (LASIK) or photorefractive keratectomy (PRK) performed within one year prior to Screening and throughout the study period.
13. Ophthalmic artificial tear drop use within 2 hours prior to any study visit. Any OTC artificial tear (preserved or unpreserved) should be continued at the same frequency and with no change in drop brand.
14. Contact lens wear within 12 hours prior to Screening or any study visit; subjects determined to have worn contact lenses within 12 hours must be rescheduled.
15. History of cauterization of the punctum or existing silicone punctal plug(s); history of silicone plug removal or collagen plug insertion or removal within 12 months prior to Screening and throughout the study period.
16. Started or changed the dose of systemic medications known to affect tear production within 30 days prior to Screening and throughout the study period. Short-term, as-needed dosing of a systemic medication is allowed with certain restrictions. One 7-day course of systemic antihistamines is allowed, but not within 7 days of Screening or any other study visit. One short (≤ 72 hour) course of the other systemic medications that affect tear production is allowed but not within 30 days of Screening or on the day of any other study visit. These include, but are not limited to, the following medications:

    * Immunomodulators
    * Tricyclic antidepressants
    * Diuretics
    * Corticosteroids (intranasal, inhaled, topical dermatological, and perianal steroids are permitted)
17. Use of any topical prescription ophthalmic medications (including cyclosporine [Restasis®, Cequa®] or topical lifitegrast [Xiidra®], steroids, nonsteroidal anti-inflammatory drugs [NSAIDs], anti-glaucoma medications, anti-microbials), topical macrolides, or oral nutraceuticals (fish, flax, black currant seed oils, etc.) within 21 days prior to Screening and throughout the study period.
18. Use of oral tetracyclines or oral macrolides within 21 days prior to Screening and throughout the study period; use of isotretinoin (Accutane®) within 90 days prior to Screening and throughout the study period.
19. Chronic daily use (defined as > 7 consecutive days at the recommended dosing frequency) of oral NSAIDs during the study period. ANY use of oral NSAIDs during the study period must be discussed with the Medical Monitor. Aspirin of any dosage is permitted.
20. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. Acceptable methods include the use of at least one of the following: intrauterine device (IUD), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence. An adult woman is considered to be of childbearing potential unless she is 1 year postmenopausal or postsurgical hysterectomy. All women of childbearing potential, including those post-tubal ligation, must have a negative urine pregnancy test result at Visit 1 (Screening), Visit 2 (Baseline), and Visit 4 (Day 84) examinations and must intend to not become pregnant during the study.
21. Participation in any drug or device clinical investigation within 30 days prior to entry into this study and/or during the period of study participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Eye Research Foundation, Newport Beach, California
  - Michael K Tran Inc, Westminster, California
  - Shettle Eye Research inc, Largo, Florida
  - Clayton Eye Clinical Research, Morrow, Georgia
  - Kannarr Eye Care, Pittsburg, Kansas
  - Heart of America Eye Care, Shawnee Mission, Kansas
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Silverstein Eye Centers, Kansas City, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Abrams Eye Center, Cleveland, Ohio
  - West Bay Eye Associates, Warwick, Rhode Island
  - Total Eye Care, Memphis, Tennessee
  - Advancing Vision Research, Nashville, Tennessee
  - R and R Eye Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OmegaD: OmegaD Softgels
  Omega 3 fatty acid Softgels. 4 Softgels administered daily at bedtime
- Placebo: Placebo Softgels
  Mineral oil Softgels, 4 Softgels administered daily at bedtime
Period: Overall Study
Arm/Group | OmegaD | Placebo
Started | 157 | 165
Completed | 157 | 165
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OmegaD | Placebo | Total
Number analyzed (Participants) | 157 | 165 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (13.4) | 56.5 (14.0) | 57.0 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 140 | 268
  Male | 29 | 25 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 11 | 19
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 37 | 36 | 73
  White | 109 | 118 | 227
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 157 | 165 | 322

OUTCOME MEASURES:

1. Primary Outcome: Tear Osmolarity
Description: Mean change from baseline in tear osmolarity to Day 84 in the study eye. One eye (the designated study eye) was was analyzed for each participant. Lower values in tear osmolarity are considered to be better, therefore the larger the number for the change from baseline to Day 84 is considered to be better.
Time Frame: 84 days
Population: Mean change from baseline to Day 84
Measure: Mean (Standard Deviation); unit: mOsm/L
Units Other Than Participants: Eyes
Arm/Group | OmegaD | Placebo
Number analyzed (Participants) | 150 | 159
Number analyzed (Eyes) | 150 | 159
mOsm/L | 13.4 (17.1) | 11.8 (13.2)

2. Primary Outcome: Ocular Surface Disease Index (OSDI)
Description: Mean change from baseline in OSDI to Day 84 in the study eye. One eye (the designated study eye) was was analyzed for each participant. The OSDI is a patient reported outcome measured on a scale from 0 to 100 where higher scores represent greater disability. The overall score is calculated using a chart based on the sum of patient responses to 12 questions each rated on a scale from 0 to 4 where higher scores represent worse outcomes.
Time Frame: 84 days
Population: Mean change from baseline to Day 84
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | OmegaD | Placebo
Number analyzed (Participants) | 151 | 162
Number analyzed (Eyes) | 151 | 162
score on a scale | 19.9 (20.1) | 19.4 (18.5)

3. Secondary Outcome: Tear Break Up Time (TBUT)
Description: Mean change from baseline in TBUT to Day 84 in the study eye. One eye (the designated study eye) was was analyzed for each participant. TBUT is measured as the number of seconds the tear film takes to break up following administration of a drop of fluorescein dye to the eye. Longer times (higher values) represent better outcomes.
Time Frame: 84 days
Population: Mean change from baseline to Day 84
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Eyes
Arm/Group | OmegaD | Placebo
Number analyzed (Participants) | 150 | 159
Number analyzed (Eyes) | 150 | 159
Seconds | 0.6 (1.7) | 0.6 (1.9)

4. Secondary Outcome: Schirmers Test
Description: Mean change from baseline in Schirmers Test to Day 84 in the study eye. One eye (the designated study eye) was was analyzed for each participant. The test measures the distance in mm that tears travel along the Schirmer test strip (filter strip) after 5 minutes following the placement of the strip in the eye. Higher values represent better outcomes.
Time Frame: 84 days
Population: Mean change from baseline to Day 84
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | OmegaD | Placebo
Number analyzed (Participants) | 150 | 159
Number analyzed (Eyes) | 150 | 159
mm | 1.13 (6.99) | 0.53 (6.34)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | OmegaD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/165
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/165
Other Adverse Events (participants affected / at risk) | 17/157 | 17/165
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OmegaD (N=157) | Placebo (N=165)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 6 (6)
Conjunctival hyperemia (Eye disorders) | 3 (3) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastroenteritis viral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Insomnia (Nervous system disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT04181593/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT04181593/SAP_001.pdf